CLINICAL TRIAL: NCT01510093
Title: Interactions Between Exogenous Insulin Aspart, Endogenous Insulin and Plasma Glucose in Type 2 Diabetes Mellitus Patients
Brief Title: Diurnal Variation of Exogenous Peptides (Endogenous Insulin Jurgita II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jurgita Janukonyte, Medical doctor, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1811
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus, endogenous insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Aspart without glucose supply (Other): Treatment with continuous subcutaneous Insulin Aspart 0.5-1.5 IE/time infusion overnight without intravenous glucose supply
  Interventions: Drug: Insulin Aspart 100 IE/ml
- Insulin Aspart with glucose supply (Other): Treatment with continuous subcutaneous Insulin Aspart 0.5-1.5 IE/time infusion overnight combined with intravenous glucose supply
  Interventions: Drug: Insulin Aspart 100 IE/ml

INTERVENTIONS:
Drug: Insulin Aspart 100 IE/ml — 1.5 IE/hour/subject/visit. Each vist takes 10 hours
  Other Names: NovoRapid 100 IE/ml

SUMMARY:
This is an exploratory trial with two cross-over arms investigating pharmacokinetic profiles of endogenous and exogenous insulin in type 2 diabetes mellitus patients treated with continuous subcutaneous Insulin Aspart infusion and combined with or without intravenous glucose infusion. The order of treatment session will be randomised.

Hypotheses:

1. Secretion of endogenous insulin depends on exogenous insulin supply
2. Secretion of endogenous insulin is depends on plasma glucose levels

DETAILED DESCRIPTION:
There are a screening visit and two treatment sessions:

Session A: Treatment with Insulin Aspart 1.5 IE/time overnight without intravenous glucose infusion Session B: Treatment with Insulin Aspart 1.5 IE/time overnight with intravenous glucose infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* Insulin-naive patients
* HbA1C < 9%
* Women and men >= 35 and <= 75 years old
* BMI 25-42 kg/m2, both values are included

Exclusion Criteria:

* Suspected or known allergy to the trial drug or similar medications
* Treatment with hte drugs that after Investigator judgment could potentially interfere with plasma glucose levels
* Heart: Unstable angina pectoris, acute myocardial infarction within the last 12 months
* Severe uncontrolled hypertension with blood pressure in lying position > 180/110 mmHg
* Impaired liver function with liver parameters more than 2 times above the upper normal limit according to the local laboratory
* Impaired kidney function with eGFR < 50 ml/min according to the local laboratory
* Pregnancy, lactation or desire for pregnancy in the study period and for women in childbearing age without adequate contraception-adequate contraception is: sterilisation, hysterectomy or current use of contraceptive pills, coil, gestagen depot injection, subdermal implantation, hormonal vaginal ring and transdermal depot patch.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profiles of endogenous insulin and Insulin Aspart | 10 hours
  Pharmacokinetic profiles of endogenous insulin and Insulin Aspart in type 2 diabetes melitus patients treated with continuous subcutaneous Insulin Aspart infusion by insulin pump and combined with or without intravenous supply of glucose

SECONDARY OUTCOMES:
Pharmacodynamic glucose profiles | 10 hours
  Pharmacodynamic glucose profiles after treatment with Insulin Aspart administred by insulin pump as a continuous subcutaneous infusion .

CONTACTS AND LOCATIONS:
Overall Officials: Jurgita Janukonyte, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of Endocrinology and Internal Diseases, Aarhus C, Central Jutland, Denmark

REFERENCES:
- [Derived] Janukonyte J, Parkner T, Bruun NH, Lauritzen T, Christiansen JS, Laursen T. Interaction between exogenous insulin, endogenous insulin, and glucose in type 2 diabetes patients. Diabetes Technol Ther. 2015 May;17(5):335-42. doi: 10.1089/dia.2014.0326. Epub 2015 Mar 18. PMID 25785658